CLINICAL TRIAL: NCT01476839
Title: Phase I Study of Yttrium-90 Labeled Anti-CD25 (a-Tac) Monoclonal Antibody Plus BEAM for Autologous Hematopoietic Cell Transplantation (AHCT) in Patients With Primary Refractory or Relapsed Hodgkin Lymphoma, the "a-Tac BEAM Regimen"
Brief Title: Radiolabeled Monoclonal Antibody Therapy and Combination Chemotherapy Before Stem Cell Transplant in Treating Patients With Primary Refractory or Relapsed Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08179; NCI-2011-03334 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA030206 (NIH); R21CA185875-01 (NIH)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Adult Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Basiliximab; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiolabeled monoclonal antibody, chemotherapy) (Experimental): DOSIMETRY STUDY: Patients receive basiliximab IV and indium In 111 basiliximab IV on day -21. Patients undergo indium In 111 imaging scans daily. Patients with appropriate biodistribution continue on to treatment.
  TREATMENT: Patients receive basiliximab IV and yttrium Y 90 basiliximab IV on day -14. Patients also receive BEAM chemotherapy comprising carmustine IV over 2 hours on days -7 and -6, etoposide IV BID over 4 hours and cytarabine IV over 2 hours BID on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous hematopoietic progenitor cell infusion on day 0.
  Interventions: Biological: basiliximab; Drug: carmustine; Drug: etoposide; Drug: cytarabine; Drug: melphalan; Other: pharmacological study; Other: laboratory biomarker analysis; Procedure: autologous hematopoietic stem cell transplantation; Biological: yttrium Y 90-labeled basiliximab

INTERVENTIONS:
Biological: basiliximab — Given IV
  Other Names: SDZ-CHI-621; Simulect
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous hematopoietic progenitor cell infusion
Biological: yttrium Y 90-labeled basiliximab — Given IV
  Other Names: 90Y basiliximab

SUMMARY:
This phase I clinical trial studies the side effects and best dose of radiolabeled monoclonal antibody therapy when given together with combination chemotherapy before stem cell transplant and to see how well it works in treating patients with primary refractory (did not respond to treatment) or relapsed (returned after treatment) Hodgkin lymphoma. Radiolabeled monoclonal antibodies can find cancer cells and carry cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as carmustine, etoposide, cytarabine, and melphalan (BEAM), work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or stopping them from spreading. Giving radiolabeled monoclonal antibody therapy together with combination chemotherapy may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of the autologous hematopoietic cell transplantation (AHCT) regimen of yttrium Y-90 basiliximab/DOTA, given in combination with standard dose(s) of BEAM in patients with primary progressive or relapsed Hodgkin lymphoma (HL).

II. To determine the recommended phase II dose (RP2D) and characterize toxicities at each dose level - including time course.

III. To evaluate hematological recovery in terms of neutrophil and platelet engraftment time.

IV. To estimate overall response rate (ORR: complete remission [CR] + partial remission [PR]), response duration, overall survival, progression-free survival, and the cumulative incidence of non-relapse mortality and relapse/progression.

V. To estimate the radiation doses to the whole body and normal organs through serial imaging studies.

VI. To define biodistribution/extended pharmacokinetics of 111indium (In)-basiliximab/DOTA and 90Y- basiliximab/DOTA including terminal elimination, serum half-life (t1/2), and area under the curve (AUC).

OUTLINE: DOSIMETRY STUDY: Patients receive basiliximab intravenously (IV) and indium In 111 basiliximab IV on day -21. Patients undergo indium In 111 imaging scans daily. Patients with appropriate biodistribution continue on to treatment.

TREATMENT: Patients receive basiliximab IV and yttrium Y 90 basiliximab IV on day -14. Patients also receive BEAM chemotherapy comprising carmustine IV over 2 hours on days -7 and -6, etoposide IV over 4 hours twice daily (BID) and cytarabine IV over 2 hours BID on days -5 to -2, and melphalan IV on day -1. Patients undergo autologous hematopoietic progenitor cell infusion on day 0.

After completion of study treatment, patients are followed up at day 90-100, 180, 1 year, 1.5 years, and 2-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmation of HL with City of Hope (COH) pathology review
* Hodgkin lymphoma that is:

  * PIF (primary induction failure): did not enter complete remission with first line of therapy; Note: a patient with PIF who responds to salvage therapy with a PR or CR is also eligible (and would be considered PIF-sensitive)
  * Early 1st relapse: initial CR of > 3 months and < 12 months after 1st line chemotherapy
  * 1st relapsed HL in a patient who is not in CR after 2 cycles of salvage therapy
  * In 2nd or subsequent relapse (RL) whether in CR or not after salvage therapy
* Relapse/persistent disease evidenced by a computed tomography and fluorodeoxyglucose (FDG)-positron emission tomography (PET), or bone marrow biopsy
* Cardiac ejection fraction of >= 50% by echocardiogram or multi gated acquisition scan (MUGA)
* Forced expiratory volume in one second (FEV1) > 65% of predicted measured, or diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% of predicted measured
* Bilirubin =< 1.5 x normal
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) =< 2 x normal except in cases where abnormal liver function tests (LFTS) are due to involvement with HL
* Serum creatinine of =< 1.5 mg/dL, and a measured creatinine clearance of >= 60 mL/min
* Karnofsky status >= 70%
* Life expectancy >= 6 months
* Females must not be pregnant or breast feeding, and must use accepted birth control methods; males must use accepted birth control methods
* Capability of providing informed consent
* Patients will be enrolled after receiving at least two cycles of salvage cytoreductive chemotherapy and collection of at least 3.0 x 10^6 CD34 cells/kg of autologous hematopoietic progenitor cells (HPC-A) by apheresis; a minimum of 2 collection procedures is required, unless collection on day #1 > 5.0 x 10^6 CD34 cells/kg; a maximum of 10 collections is allowed; bone marrow harvest to supplement apheresis is not allowed
* Co-enrollment on Institutional Review Board (IRB) #98117, entitled Molecular Pathogenesis of Therapy-Related Leukemia
* All pre-study and follow-up imaging studies preferably performed at City of Hope
* Recovery from non-hematologic toxicities of salvage cytoreductive chemotherapy to =< grade 2 (Common Terminology Criteria for Adverse Events version 4 [CTCAE v4])
* Body mass index (BMI) > 30% will be considered on a case-by-case basis by the radiation oncology principal investigator (PI)
* While on this study, patients may not be treated with any other investigational agent for any purpose until relapse or progression

Exclusion Criteria:

* Lymphocyte-predominant Hodgkin lymphoma
* Prior high dose chemotherapy with autologous stem cell transplant, or prior allogeneic transplantation
* Significant prior external beam dose-limiting radiation to a critical organ based on review of the prior radiation treatment records by the radiation oncology PI; patients who have had prior external beam radiation > 2000 cGy (at 180 to 200 cGy per day) to any portion of the lung will be ineligible; patients with ANY prior radiation to the heart are ineligible; patients with > 500 cGy to any portion of the kidney will be excluded from the study
* Presence of antibody against basiliximab (only required for patients who have received prior antibody)
* Myelodysplasia or any active malignancy other than HL, or < 5 years remission from any other prior malignancy, except adequately treated basal cell or squamous cell carcinoma
* Active hepatitis B or C viral infection or hepatitis B surface antigen positive
* Positive human immunodeficiency virus antibody
* Patients with psychosocial circumstances or illnesses that preclude protocol participation (to be determined by PI)
* Co-morbid illnesses that preclude protocol participation (to be determined by PI)
* Any cytogenetic abnormality in the bone marrow that is known to be associated with or predictive of myelodysplasia is excluded. This includes, but is not limited to, del(5), del(7), del(11)
* Persistent marrow involvement (> 10%) with HL after salvage cytoreductive therapy and before stem cell mobilization
* Systemic chemotherapy or radiation within 4 weeks prior to the Y-90 dose of radioimmunotherapy (RIT), with the exception of single agent Cytoxan priming chemotherapy administered for mobilization
* Bone marrow (BM) harvest required to reach adequate cell dose for transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
RP2D of Yttrium-90 labeled basiliximab | Up to 18 months
  RP2D will generally be the highest maximum tolerated dose (MTD), but it may be less than the MTD based on a review of available data/cumulative toxicities. Additional pulmonary toxicity monitoring will be performed among enrolled/treated patients with prior brentuximab vedotin exposure for both portions of the study.
DLT | For 30 days post-transplant
  Toxicities will be recorded using two distinct grading systems: the modified Bearman Scale and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.0 scale. Observed toxicities will be summarized by type, severity, date of onset, duration (for neutropenia only), and attribution.

SECONDARY OUTCOMES:
Best ORR | Up to 5 years
  Response will be evaluated using the revised Cheson criteria. Objective tumor response for all patients will be summarized for each dose level, and the number and percent responding combined across dose levels.
Biodistribution of basiliximab | Pre-basiliximab infusion; pre radiolabeled basiliximab infusion; 2 and 4-6 hours post radiolabeled basiliximab infusion; and then 1, 2, 3-4, 5, and 6 days post radiolabeled basiliximab infusion
  Serum basiliximab levels will be evaluated. T1/2 and alpha- and beta- phase will be estimated for each patient using compartmental and non-compartmental methods, with summary statistics tabulated. Exploratory models to predict tumor response, survival, and toxicities from serum data and patient characteristics will be performed to better understand the effect of treatment on patients.
Cumulative incidence of non-relapsed mortality (NRM) | From stem cell infusion to death from any cause other than disease relapse or progression, assessed up to 5 years
  Cumulative relapse incidence will be estimated treating non-relapse related death events as competing risks and conversely, NRM will be calculated controlling for relapse as a competing risk. Cumulative incidence of NRM and relapse-related mortality will be calculated using the method of Gooley et al. Cumulative incidence differences will be assessed by Gray's test.
Cumulative incidence of relapse/progression incidence | Up to 5 years
  Cumulative relapse incidence will be estimated treating non-relapse related death events as competing risks and conversely, NRM will be calculated controlling for relapse as a competing risk. Cumulative incidence of NRM and relapse-related mortality will be calculated using the method of Gooley et al. Cumulative incidence differences will be assessed by Gray's test.
Incidence of toxicity | Up to 100 days post-infusion
  Observed toxicities will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE v4.0 and nadir or maximum values for lab measures), dates of onset, duration, reversibility, and attribution.
Overall survival (OS) | Time from transplant to death from any cause, assessed up to 5 years
  OS will be estimated using the KM product-limit method; 95% CIs will be calculated using the logit transformation and the Greenwood variance estimate. OS will be estimated using two different start times (from radio-labeled therapeutic infusion and from stem cell infusion) to death from any cause.
Progression free survival (PFS) | Time from transplant to the first observation of disease progression or death from any cause, whichever occurs first, assessed at 5 years
  PFS will be estimated using the Kaplan-Meier (KM) product-limit method. 95% confidence intervals (CIs) will be calculated using the logit transformation and the Greenwood variance estimate. PFS will be estimated using two different start times (from radio-labeled therapeutic infusion and from stem cell infusion) to recurrence, progression, or death from any cause.
Response duration | Time from when criteria for response (CR or PR) are met to the first documentation of relapse or progression, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Smith, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Herrera AF, Palmer J, Adhikarla V, Yamauchi D, Poku EK, Bading J, Yazaki P, Dandapani S, Mei M, Chen R, Cao T, Karras N, McTague P, Nademanee A, Popplewell L, Sahebi F, Shively JE, Simpson J, Smith DL, Song J, Spielberger R, Tsai NC, Thomas SH, Forman SJ, Colcher D, Wu AM, Wong J, Smith E. Anti-CD25 radioimmunotherapy with BEAM autologous hematopoietic cell transplantation conditioning in Hodgkin lymphoma. Blood Adv. 2021 Dec 14;5(23):5300-5311. doi: 10.1182/bloodadvances.2021004981. PMID 34638132